CLINICAL TRIAL: NCT04120389
Title: Efficacy of an Ocular Bandage Contact Lens for the Treatment of Dry Eye After Complicated and Combined Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xuwen2019-929
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-01

CONDITIONS: Cataract; Lens Subluxation; Hypermature Cataract; Corneal Opacity; Small Pupil
Keywords: Bandage contact lens; cataract surgery; dry eye
MeSH Terms: conditions — Cataract; Lens Subluxation; Corneal Opacity; Miosis; Dry Eye Syndromes | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCL group (Experimental): bandage contact lenses(PureVision; Bausch & Lomb Inc., Rochester, NY)
  Interventions: Device: bandage contact lenses(PureVision; Bausch & Lomb Inc., Rochester, NY); Procedure: phacoemulsification
- control group (Active Comparator)
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Device: bandage contact lenses(PureVision; Bausch & Lomb Inc., Rochester, NY) — wear an bandage contact lenses for a week after Complicated and Combined cataract surgery.
  Arms: BCL group
Procedure: phacoemulsification — underwent standard phacoemulsification through a 2.8-mm clear corneal temporal incision and intraocular lens

SUMMARY:
To study the efficacy of an ocular bandage contact lens for the treatment of dry eye after complicated and combined cataract surgery

ELIGIBILITY:
Inclusion Criteria:

1. cataract patients（age 40-80）
2. complex symptom（such as:corneal opacity、small pupil、zonule relaxationlens subluxation、Shallow Anterior Chamber、hypermature cataract、hard nucleus,etc）
3. dry eye disease

Exclusion Criteria:

1. simplex age-related cataract
2. contact lens use
3. ocular therapies such as 0.05% cyclosporine A or steroids in the last 3 months
4. any systemic diseases such as heart diseases, diabetes and psychosis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index questionnaire | 0 day preoperatively
  Ocular Surface Disease Index questionnaire were included 12 questions，and each was rated from 0-4
Ocular Surface Disease Index questionnaire | 1 day postoperatively
  Ocular Surface Disease Index questionnaire were included 12 questions，and each was rated from 0-4
Ocular Surface Disease Index questionnaire | 1 week postoperatively
  Ocular Surface Disease Index questionnaire were included 12 questions，and each was rated from 0-4
Ocular Surface Disease Index questionnaire | 1 month postoperatively
  Ocular Surface Disease Index questionnaire were included 12 questions，and each was rated from 0-4
Ocular Surface Disease Index questionnaire | 3 months postoperatively
  Ocular Surface Disease Index questionnaire were included 12 questions，and each was rated from 0-4
Tear Breakup Time | 0 day preoperatively
  Tear Breakup Time was performed to assess tear film stability
Tear Breakup Time | 1 week postoperatively
  Tear Breakup Time was performed to assess tear film stability
Tear Breakup Time | 1 month postoperatively
  Tear Breakup Time was performed to assess tear film stability
Tear Breakup Time | 3 months postoperatively
  Tear Breakup Time was performed to assess tear film stability
Schirmer test with anesthesia | 0 day preoperatively
  The Schirmer test was performed by inserting a test strip
Schirmer test with anesthesia | 1 week postoperatively
  The Schirmer test was performed by inserting a test strip
Schirmer test with anesthesia | 1 month postoperatively
  The Schirmer test was performed by inserting a test strip
Schirmer test with anesthesia | 3 months postoperatively
  The Schirmer test was performed by inserting a test strip

SECONDARY OUTCOMES:
Subjective symptoms | 0 day preoperatively
  Subjective symptoms evaluation related to 11 ocular symptoms ，and each was graded as follows：0 never、1 occasional、2 often、3 always
Subjective symptoms | 1 day postoperatively
  Subjective symptoms evaluation related to 11 ocular symptoms ，and each was graded as follows：0 never、1 occasional、2 often、3 always
Subjective symptoms | 1 week postoperatively
  Subjective symptoms evaluation related to 11 ocular symptoms ，and each was graded as follows：0 never、1 occasional、2 often、3 always
Subjective symptoms | 1 month postoperatively
  Subjective symptoms evaluation related to 11 ocular symptoms ，and each was graded as follows：0 never、1 occasional、2 often、3 always
Subjective symptoms | 3 months postoperatively
  Subjective symptoms evaluation related to 11 ocular symptoms ，and each was graded as follows：0 never、1 occasional、2 often、3 always
Fluorescein Staining | 0 day preoperatively
  The corneal surface was divided into four regions, and each region was scored as follows: 0, no staining; 1, between one and three dots; 2, less than five dots; and 3, bulk or strip staining. The four regions scores were then added to obtain a final score for the eye
Fluorescein Staining | 1 week postoperatively
  The corneal surface was divided into four regions, and each region was scored as follows: 0, no staining; 1, between one and three dots; 2, less than five dots; and 3, bulk or strip staining. The four regions scores were then added to obtain a final score for the eye
Fluorescein Staining | 1 month postoperatively
  The corneal surface was divided into four regions, and each region was scored as follows: 0, no staining; 1, between one and three dots; 2, less than five dots; and 3, bulk or strip staining. The four regions scores were then added to obtain a final score for the eye
Fluorescein Staining | 3 months postoperatively
  The corneal surface was divided into four regions, and each region was scored as follows: 0, no staining; 1, between one and three dots; 2, less than five dots; and 3, bulk or strip staining. The four regions scores were then added to obtain a final score for the eye

OTHER OUTCOMES:
Best Corrected Visual Acuity | 0 day preoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 1 day postoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 1 week postoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 1 month postoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 3 months postoperatively
  The BCVA was measured by the same optometrist at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen D, Xu D, Wu X, Wang J, Sheng S, Yu X, Lin X, Liu L, Ge X, Zhao H, Xu W. The efficacy of bandage contact lens in relieving the aggravation of dry eye disease after complicated cataract or/and IOL surgery. BMC Ophthalmol. 2024 Mar 28;24(1):141. doi: 10.1186/s12886-024-03385-x. PMID 38549070